CLINICAL TRIAL: NCT00254683
Title: Study of the Value of the PET/CT in Evaluating the Response of Distal Rectal Cancer to Neoadjuvant Chemoradiation Therapy
Brief Title: Use of Positron Emission Tomography/Computed Tomography (PET/CT) to Assess Tumor Response to Neoadjuvant Treatment for Distal Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rodrigo Oliva Perez, University of São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 717/05
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Positron Emission Tomography; Fluorodeoxyglucose F18; Computed Tomography; Neoadjuvant Therapy; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/CT (Experimental): Single arm study evaluating the use of PET/CT to assess rectal cancer response to neoadjuvant therapy
  Interventions: Device: PET/CT with FDG

INTERVENTIONS:
Device: PET/CT with FDG — PET/CT before start of neoadjuvant CRT, at 6 weeks, 12 weeks, following CRT completion and 12mo, 24mo following CRT for those considered complete responders
  Other Names: PET-CT

SUMMARY:
Preoperative chemoradiation therapy is the preferred initial treatment option for distal rectal cancers. However, assessing tumor response to preoperative chemoradiation therapy remains a challenge to the colorectal surgeon, especially when determining if there is a complete response, observed in more than 10% of cases. The purpose of this study is to evaluate the use of the PET/CT in assessing distal rectal tumor response to preoperative chemoradiation therapy.

DETAILED DESCRIPTION:
Patients with distal rectal adenocarcinoma will be submitted to an initial whole body PET/CT prior to the preoperative chemoradiation therapy with 5-fluorouracil and 5040 cGy. Six weeks and 12 weeks after the preoperative treatment is finished the PET/CT will be repeated. At 1 and at 2 years after preoperative treatment is concluded another PET/CT will be performed. The colorectal surgeon evaluating the response to chemoradiation therapy will be blinded to the results of the PET/CT, as the radiologist will be blinded to the response assessment. PET/CT results will not be used to determine treatment strategy, unless metastatic disease or other disease is diagnosed. Patients with a complete clinical response at 8 weeks will be rigorously followed while patients with an incomplete clinical response at 8 weeks will be submitted to radical surgery. PET/CT results will be compared to current radiological studies and final pathological reports.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rectal Adenocarcinoma
* Location of Tumor less than 7cm from Anal Verge

Exclusion Criteria:

* Pregnancy or Nursing
* Metastatic Disease (Stage IV disease)
* Previous treatment for any cancer
* Patients clinically unable to receive neoadjuvant chemoradiotherapy
* Hypersensitivity to 18FDG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Primary Completion 2010-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
PET/CT specificity and sensitivity for tumor response | Response assesment at 6 and 8 weeks following neoadjuvant therapy

SECONDARY OUTCOMES:
Correlation between PET/CT and complete clinical Response | 2 years following completion of neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Angelita Habr-Gama, MD, PhD, Study Director — University of São Paulo School of Medicine - Department of Gastroenterology; Rodrigo O Perez, MD, Principal Investigator — University of São Paulo School of Medicine - Department of Gastroenterology; Joaquim J Gama-Rodrigues, MD, PhD, Study Chair — University of São Paulo School of Medicine - Department of Gastroenterology; Carlos A Buchpiguel, MD, PhD, Principal Investigator — University of São Paulo School of Medicine - Department of Radiology; Desedério R Kiss, MD, PhD, Principal Investigator — University of São Paulo School of Medicine - Department of Gastroenterology
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Habr-Gama A, Perez RO, Sao Juliao GP, Proscurshim I, Fernandez LM, Figueiredo MN, Gama-Rodrigues J, Buchpiguel CA. Consolidation chemotherapy during neoadjuvant chemoradiation (CRT) for distal rectal cancer leads to sustained decrease in tumor metabolism when compared to standard CRT regimen. Radiat Oncol. 2016 Feb 24;11:24. doi: 10.1186/s13014-016-0598-6. PMID 26911200
- [Derived] Perez RO, Habr-Gama A, Sao Juliao GP, Lynn PB, Sabbagh C, Proscurshim I, Campos FG, Gama-Rodrigues J, Nahas SC, Buchpiguel CA. Predicting complete response to neoadjuvant CRT for distal rectal cancer using sequential PET/CT imaging. Tech Coloproctol. 2014 Aug;18(8):699-708. doi: 10.1007/s10151-013-1113-9. Epub 2014 Feb 8. PMID 24509716
- [Derived] Perez RO, Habr-Gama A, Sao Juliao GP, Gama-Rodrigues J, Sousa AH Jr, Campos FG, Imperiale AR, Lynn PB, Proscurshim I, Nahas SC, Ono CR, Buchpiguel CA. Optimal timing for assessment of tumor response to neoadjuvant chemoradiation in patients with rectal cancer: do all patients benefit from waiting longer than 6 weeks? Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1159-65. doi: 10.1016/j.ijrobp.2012.01.096. Epub 2012 May 12. PMID 22580120
- [Derived] Perez RO, Habr-Gama A, Gama-Rodrigues J, Proscurshim I, Juliao GP, Lynn P, Ono CR, Campos FG, Silva e Sousa AH Jr, Imperiale AR, Nahas SC, Buchpiguel CA. Accuracy of positron emission tomography/computed tomography and clinical assessment in the detection of complete rectal tumor regression after neoadjuvant chemoradiation: long-term results of a prospective trial (National Clinical Trial 00254683). Cancer. 2012 Jul 15;118(14):3501-11. doi: 10.1002/cncr.26644. Epub 2011 Nov 15. PMID 22086847